CLINICAL TRIAL: NCT04416009
Title: the Determination of Extracellular Water (ECW) Which is Detected by Bioimpedence Method on Severe and Mild Covid 19 Pneumonia Clinical Course
Brief Title: Extracellular Water in Covid 19 Pneumonia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Gaziosmanpasa Research and Education Hospital (Other Government)
Responsible Party: Principal Investigator, SİBEL BEKTAŞ, director, Gaziosmanpasa Research and Education Hospital
Other Study IDs: 76
Record Dates: First submitted 2020-06-01; First posted 2020-06-04 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-06

CONDITIONS: Extracellular Fluid Alteration; Corona Virus Infection
Keywords: covid-19; NİCaS; pneumonia
MeSH Terms: conditions — Coronavirus Infections; COVID-19; Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- mild pneumonia ECW: the covid 19 pneumonia patients who hospitalised to the ward
  Interventions: Device: NİCaS
- severe pneumonia ECW: the covid 19 pneumonia patients who hospitalised to the intensive care unit
  Interventions: Device: NİCaS

INTERVENTIONS:
Device: NİCaS — whole body bioimpedence method

SUMMARY:
According to various studies Covid 19 pneumonia has a very similar clinical course to Acute Respiratory Distress Syndrome (ARDS) which has clarified by Berlin definition. Based on this similarity, extracellular fluid of lungs and diffuse alveolar damage should be observed in covid 19 pneumonia as well. Extracellular water (ECW) can be determine by using whole body bioimpedence system (NİCaS). The aim of this study is to investigate the effect of ECW on the clinical apperence of covid 19 pneumonia clinical course.

DETAILED DESCRIPTION:
Increase in the extracellular water of lungs is the major pathophisilogy of ARDS. According to various studies Covid 19 pneumonia has a very similar clinical course to Acute Respiratory Distress Syndrome (ARDS) which has clarified by Berlin definition. Depending on the similarity of Covid 19 and ARDS; evaluation of ECW ,can be a determinant of clinical apperence of covid19 pneumonia. The aim of this study to find the corelation between ECW and severty of the pneumonia.

In this prospective -controlled research, the patients who were diagnosed with Covid-19 pneumonia will be evaluated. The ones in the intensive care will be considered as severe, and the ones in the ward will be considered as mild clinical course pneumonia. İn both groups, in addition to other heamodynamic parametres, ECW will be recorded using non-invasive body biooimpedence method by NİCaS machine. The total amount of patients will be 52, 26 each two groups.

The ward and intensive care patients will be connected to the NİCaS machine to determine ECW and statistically significantchanges will be recorded. The device consists of a laptop, a software which calculates cardiac parameters and two electrodes. The measurement is done by the following process: one of these electrodes, which looks like ECG electrodes, is stuck to the wrist and the other one to the opposite ankle or each one to two wrists.

the severety of illness will try to be detected.Gpower 3 for Mac Os (Faul, F., Erdfelder, E., Buchner, A., & Lang, A.-G. (2009). Statistical power analyses using G*Power 3.1: Tests for correlation and regression analyses. Behavior Research Methods, 41, 11491160.) was used for istatistical power analysis.The power analysis was done priorly and based on the T-test.In order to provide enoughsample magnitude power, which is 0.8, it was calculated that each group should have 26 patients which makes at total of 52 Statistical method: The normal distribution of data will be evaluated using Kolmogorov-Smirnov test. Parametric ones will be used in normal distrubitions, non-parametric ones will be used in abnormal distrubitions. İntergroup ECW values will be compared via independent sample T test. In catagoric data, the comparisons will be made with Pearson Ki square test, and the p values less then 0.05 will be considered as significant.

ELIGIBILITY:
Inclusion Criteria:

Covid 19 pneumonia, hospitalized patients older than 18

Exclusion Criteria:

younger than 18 years old, patients not infected with covid 19

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospitalized covid 19 patients
Sampling Method: Probability Sample
Enrollment: 52 (Estimated)
Dates: Start 2020-07-05 (Estimated); Primary Completion 2020-12-20 (Estimated); Study Completion 2021-02-20 (Estimated)

PRIMARY OUTCOMES:
ECW | three measurements with half an hour intervals
  Changes of three measurements of extracellular water in both lungs

CONTACTS AND LOCATIONS:
Locations (1):
- Gaziosmanpaşa TREH, Istanbul, Gaziosmanpaşa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tagami T, Ong MEH. Extravascular lung water measurements in acute respiratory distress syndrome: why, how, and when? Curr Opin Crit Care. 2018 Jun;24(3):209-215. doi: 10.1097/MCC.0000000000000503. PMID 29608455
- [Background] Jozwiak M, Teboul JL, Monnet X. Extravascular lung water in critical care: recent advances and clinical applications. Ann Intensive Care. 2015 Dec;5(1):38. doi: 10.1186/s13613-015-0081-9. Epub 2015 Nov 6. PMID 26546321